CLINICAL TRIAL: NCT03359785
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled, Cross-Over Study to Evaluate Pharmacodynamic Effects, Safety, Tolerability, and Pharmacokinetics of Multiple Oral Doses of TAK-831 in Adult Subjects With Schizophrenia
Brief Title: A Study to Evaluate Multiple Oral Doses of Luvadaxistat in Adults With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-831-2001; 2017-001739-38 (EudraCT Number); U1111-1197-9766 (Other: World Health Organization); 17/YH/0196 (Registry Identifier: NRES)
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: Schizophrenia
Keywords: Drug therapy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Luvadaxistat 500 mg, then Placebo (Experimental): Participants first received luvadaxistat 500 mg orally once daily (QD) for 8 days during treatment period 1. After a washout of 14 to 21 days, participants then received matching placebo orally QD for 8 days during treatment period 2.
  Interventions: Drug: Luvadaxistat; Drug: Matching Placebo
- Placebo, then Luvadaxistat 500 mg (Experimental): Participants first received matching placebo orally QD for 8 days during treatment period 1. After a washout of 14 to 21 days, participants then received luvadaxistat 500 mg orally QD for 8 days during treatment period 2.
  Interventions: Drug: Luvadaxistat; Drug: Matching Placebo
- Luvadaxistat 50 mg, then Placebo (Experimental): Participants first received luvadaxistat 50 mg orally QD for 8 days during treatment period 1. After a washout of 14 to 21 days, participants then received matching placebo orally QD for 8 days during treatment period 2.
  Interventions: Drug: Luvadaxistat; Drug: Matching Placebo
- Placebo, then Luvadaxistat 50 mg (Experimental): Participants first received matching placebo orally QD for 8 days during treatment period 1. After a washout of 14 to 21 days, participants then received luvadaxistat 50 mg orally QD for 8 days during treatment period 2.
  Interventions: Drug: Luvadaxistat; Drug: Matching Placebo

INTERVENTIONS:
Drug: Luvadaxistat — TAK-831 Tablets.
  Other Names: TAK-831; NBI-1065844
Drug: Matching Placebo — Matching Placebo Tablets.

SUMMARY:
The purpose of this study is to determine whether luvadaxistat is superior to placebo in improving cerebellar function as measured with the average percentage of conditioned responses during the eyeblink conditioning (EBC) test.

DETAILED DESCRIPTION:
The drug being tested in this study is called luvadaxistat. Luvadaxistat is being tested to treat people with schizophrenia.

Participants will be randomly assigned to one of the two treatment sequences which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Luvadaxistat 500 milligrams (mg) followed by matching placebo
* Matching placebo followed by luvadaxistat 50 mg

Participants will receive luvadaxistat 500 mg during the treatment period in which they are assigned to luvadaxistat. Following an interim analysis, there will be a study-wide decision about whether to treat the additional participants with luvadaxistat 500 mg during the active treatment period to or treat them with luvadaxistat 50 mg during this period. After the interim analysis, the participant and study doctor will not be aware of which luvadaxistat dose is being used.

ELIGIBILITY:
Inclusion Criteria:

* Have a body mass index (BMI) greater than or equal to (>=) 18.5 and less than or equal to (<=) 40.0 (kilogram per square meter [kg/m^2]) at the Screening Visit.
* With a current Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of schizophrenia who are receiving stable antipsychotic therapy (no increase, no decrease greater than [>] 20% in dose in the preceding 2 months).
* Positive and Negative Syndrome Scale (PANSS) negative symptom factor score (NSFS) >= 15, stable screening and baseline PANSS NSFS (< 25% change).
* PANSS total score <= 90; stable screening and baseline PANSS total score (less than [<] 20% change).
* Receiving stable (no increase, no decrease > 25% in dose in the preceding 2 months)antipsychotic medication at doses not to exceed risperidone 6 mg or its equivalent. Concomitant treatment with a subtherapeutic dose of a second antipsychotic may be permitted with sponsor or designee approval if used as a hypnotic (maximum of quetiapine 300 mg or its equivalent once daily at bedtime) and participants does not show morning sedation as per the investigator opinion, but not if it is used for refractory positive psychosis symptoms. Under this exception, the total daily dose the second antipsychotic will not have to be included in the calculation of the 6 mg/day risperidone-equivalent limit.

Exclusion Criteria:

* Has a history of cancer (malignancy) excluding treated basal cell carcinoma or treated stage 0 (in situ) cervical carcinoma.
* Has a history of significant multiple and/or severe allergies (example [eg], food, drug, latex allergy) or has had an anaphylactic reaction or significant intolerability to prescription or nonprescription drugs or food.
* Has a QT interval with Fridericia's correction method (QTcF) > 450 milliseconds [ms] (males) or > 470 ms (females) confirmed with one repeat testing, at the Screening Visit or Check-in.
* Has a positive alcohol or drug screen for disallowed substances, including amphetamines, barbiturates, cocaine, marijuana, methadone, methamphetamine, 3,4-methylenedioxymethamphetamine, phencyclidine, or nonprescribed benzodiazepines or opiates.
* Is positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies, or has HIV by history (confirmatory testing is allowed; most sensitive test should take precedence).
* Had major surgery, donated or lost 250 milliliter [mL] of blood within 4 weeks prior to the prestudy (screening) visit.
* Has a known hypersensitivity to any component of the formulation of luvadaxistat.
* Has a history of significant skin reactions (hypersensitivity) to adhesives, metals or plastic.
* Is considered by the investigator to be at imminent risk of suicide or injury to self, others, or property, or participants who within the past year prior to Screening have attempted suicide. Participants who have positive answers on item 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS) (based on the past year) prior to randomization are excluded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CBH Health, LLC, Gaithersburg, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 10 January 2018 to 21 December 2020.
Pre-assignment Details: This 2-period cross-over study assessed the pharmacodynamic (PD) effects, safety, tolerability and pharmacokinetics (PK) of multiple oral doses of luvadaxistat given once daily (QD) in adult participants with schizophrenia. Effects of 2 dose levels of luvadaxistat (500 milligrams [mg] and 50 mg) or placebo were assessed.
Groups:
- Luvadaxistat 500 mg, Then Placebo: Participants first received luvadaxistat 500 mg orally QD for 8 days during treatment period 1. After a washout of 14 to 21 days, participants then received matching placebo orally QD for 8 days during treatment period 2.
Period: Overall Study
Arm/Group | Luvadaxistat 500 mg, Then Placebo | Placebo, Then Luvadaxistat 500 mg | Luvadaxistat 50 mg, Then Placebo | Placebo, Then Luvadaxistat 50 mg
Started | 8 | 9 | 7 | 7
Completed | 6 | 6 | 5 | 7
Not Completed | 2 | 3 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Early study termination due to study pause | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were randomized and received at least 1 dose of double-blind study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Luvadaxistat 500 mg, Then Placebo | Placebo, Then Luvadaxistat 500 mg | Luvadaxistat 50 mg, Then Placebo | Placebo, Then Luvadaxistat 50 mg | Total
Number analyzed (Participants) | 8 | 9 | 7 | 7 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 7 | 7 | 31
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 1 | 2 | 5
  Male | 8 | 7 | 6 | 5 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 9 | 6 | 7 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 8 | 6 | 4 | 26
  White | 0 | 1 | 0 | 2 | 3
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Percent of Conditioned Responses During the Eye Blink Conditioning (EBC) Test at Day 8
Description: EBC is a method used to investigate cerebellar-dependent learning. In EBC, a conditioned stimulus, a tone precedes but co-terminates with an unconditioned stimulus, an airpuff to the eyelid. Learning is demonstrated when an eyeblink (the conditioned response) occurs prior to the onset of the unconditioned stimulus. The percentage can range from 0% (no conditioned learning has occurred) to 100% (all responses are conditioned). Results are reported as least squares (LS) means at Day 8, determined using an analysis of variance (ANOVA).
Time Frame: Baseline, Day 8 of each treatment period
Population: The PD set consisted of all randomized participants who received at least 1 dose of study treatment and had at least 1 post- dose PD result. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent of Conditioned Responses
Groups:
- Luvadaxistat 50 mg: Participants received luvadaxistat 50 mg orally QD for 8 days during either treatment periods 1 or 2 of the study.
- Placebo (Reference for Luvadaxistat 50 mg): Participants received matching placebo orally QD for 8 days during either treatment periods 1 or 2 of the study. Placebo treatment in this arm corresponds to participants who received 50 mg luvadaxistat in the alternative treatment period (that is, participants receiving 50 mg and 500 mg luvadaxistat were analyzed separately and placebo treatment was not pooled).
- Luvadaxistat 500 mg: Participants received luvadaxistat 500 mg orally QD for 8 days during either treatment periods 1 or 2 of the study.
- Placebo (Reference for Luvadaxistat 500 mg): Participants received matching placebo orally QD for 8 days during either treatment periods 1 or 2 of the study. Placebo treatment in this arm corresponds to participants who received 500 mg luvadaxistat in the alternative treatment period (that is, participants receiving 50 mg and 500 mg luvadaxistat were analyzed separately and placebo treatment was not pooled).
Arm/Group | Luvadaxistat 50 mg | Placebo (Reference for Luvadaxistat 50 mg) | Luvadaxistat 500 mg | Placebo (Reference for Luvadaxistat 500 mg)
Number analyzed (Participants) | 10 | 12 | 11 | 11
Percent of Conditioned Responses | 0.597 (0.459) | 0.319 (0.432) | 0.578 (0.444) | 1.344 (0.428)
Statistical Analysis 1: Comparison: Luvadaxistat 50 mg vs Placebo (Reference for Luvadaxistat 50 mg); Test type: Superiority; p = 0.2401, ANOVA; LS Mean Difference = 0.278, 90% CI 1-sided [lower limit -0.246], Standard Error of Mean 0.376
Statistical Analysis 2: Comparison: Luvadaxistat 500 mg vs Placebo (Reference for Luvadaxistat 500 mg); Test type: Superiority; p = 0.9053, ANOVA; LS Mean Difference = -0.766, 90% CI 1-sided [lower limit -1.513], Standard Error of Mean 0.547

2. Secondary Outcome: Change From Baseline in the Mean Mismatch Negativity (MMN) at Day 8
Description: MMN is an event related potential (ERP) evoked in response to unattended changes in background stimulation. MMN reflects an automatic process of detecting a mismatch between a deviant stimulus and a sensory-memory trace. Smaller amplitudes of MMN have been consistently identified in schizophrenia participants. MMN amplitude was measured at midline frontal electrode (Fz) of electroencephalogram (EEG). Baseline was defined as the last observation prior to the dose of study treatment in the corresponding period. Results are reported as LS mean change from baseline at Day 8, determined using an ANOVA.
Time Frame: Baseline, Day 8 of each treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: microvolts
Arm/Group | Luvadaxistat 50 mg | Placebo (Reference for Luvadaxistat 50 mg) | Luvadaxistat 500 mg | Placebo (Reference for Luvadaxistat 500 mg)
Number analyzed (Participants) | 13 | 12 | 15 | 15
microvolts | -0.239 (0.363) | 0.669 (0.382) | 0.594 (0.492) | -0.154 (0.501)

3. Secondary Outcome: Change From Baseline in the Mean P300 Amplitude at Day 8
Description: The P300 wave is an ERP component that is elicited by the presentation of a novel, behaviorally relevant target stimulus embedded among irrelevant stimuli in a manner similar to MMN but requiring active listening and responding from participants. Auditory stimuli are presented in an oddball paradigm consisting of 1 standard tone and 1 target tone. Participants are instructed to push a button as quickly as possible when they hear the target tone but not when they hear the standard tone. P300 reflects allocation of attention and activation of immediate memory. P300 amplitude was measured at midline parietal electrode (Pz) of EEG. Baseline was defined as the last observation prior to the dose of study treatment in the corresponding period. Results are reported as LS mean change from baseline at Day 8, determined using an ANOVA.
Time Frame: Baseline, Day 8 of each treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: microvolts
Arm/Group | Luvadaxistat 50 mg | Placebo (Reference for Luvadaxistat 50 mg) | Luvadaxistat 500 mg | Placebo (Reference for Luvadaxistat 500 mg)
Number analyzed (Participants) | 12 | 12 | 14 | 14
microvolts | -2.019 (1.68) | 0.608 (1.68) | 1.102 (1.77) | 2.595 (1.86)

4. Secondary Outcome: Change From Baseline in the Mean Auditory Steady State Response (ASSR) at Day 8
Description: ASSRs are evoked oscillatory responses that are entrained to the frequency and phase of temporally modulated stimuli. Individuals with schizophrenia experience subjective sensory anomalies and objective deficits on assessment of sensory function. These deficits can be produced by abnormal signaling in the sensory pathways and sensory cortex or by later-stage disturbances in the cognitive processing of such inputs. ASSR can be used to assess the integrity of sensory pathways including cortical processing. The ASSR applied a frequency stimulus of 40 hertz (Hz) and was measured at midline central electrode (Cz) of EEG. Baseline was defined as the last observation prior to the dose of study treatment in the corresponding period. Results are reported as LS mean change from baseline at Day 8, determined using an ANOVA.
Time Frame: Baseline, Day 8 of each treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: microvolts-squared
Arm/Group | Luvadaxistat 50 mg | Placebo (Reference for Luvadaxistat 50 mg) | Luvadaxistat 500 mg | Placebo (Reference for Luvadaxistat 500 mg)
Number analyzed (Participants) | 13 | 12 | 15 | 14
microvolts-squared | 2.135 (8.83) | -16.282 (9.31) | 9.411 (20.4) | 9.203 (20.9)

5. Secondary Outcome: Change From Baseline on the Brief Assessment of Cognition in Schizophrenia (BACS) Composite Score at Day 7
Description: BACS is a cognition assessment battery and includes brief assessments of reasoning and problem solving, verbal fluency, attention, verbal memory, working memory and motor speed. The primary measure from each test is standardized by creating z-scores whereby the mean of the test session of a healthy person is set to 0 and the standard deviation set to 1. A Z-score of 0 represents the population mean. A composite score was calculated by averaging the 4 measures from the BACS used in the study and then calculating a z-score of the composite. The composite z-score indicates how much higher or lower the participants cognition is compared to a healthy person. Lower z-scores are indicative of lower cognitive performance. Baseline was defined as the last observation prior to the dose of study treatment in the corresponding period. Results are reported as LS mean change from baseline at Day 7, determined using an ANOVA.
Time Frame: Baseline, Day 7 of each treatment period
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Luvadaxistat 50 mg | Placebo (Reference for Luvadaxistat 50 mg) | Luvadaxistat 500 mg | Placebo (Reference for Luvadaxistat 500 mg)
Number analyzed (Participants) | 12 | 12 | 15 | 15
z-score | 2.574 (2.51) | 5.070 (2.55) | 5.696 (1.41) | -0.075 (1.43)

6. Secondary Outcome: Change From Baseline in the Mean Plasma Concentrations of D-serine and L-serine at Day 8
Description: Blood samples were collected at pre-specified timepoints and plasma concentrations of D-serine and L-serine were measured. Results are reported as LS mean change from baseline at Day 8, determined using a mixed model for repeated measures (MMRM).
Time Frame: Day 1 and at multiple time points (up to 6 hours) to Day 8 pre-dose
Population: The PK analysis set included all randomized participants who received at least 1 dose of study treatment and who had any available plasma concentration data. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mg / liter
Arm/Group | Luvadaxistat 50 mg | Placebo (Reference for Luvadaxistat 50 mg) | Luvadaxistat 500 mg | Placebo (Reference for Luvadaxistat 500 mg)
Number analyzed (Participants) | 12 | 12 | 15 | 15
mg / liter
  D-serine | 0.0402 (0.00632) | -0.000892 (0.00637) | 0.0398 (0.00710) | 0.00212 (0.00712)
  L-serine | 0.669 (0.479) | -0.543 (0.483) | -1.09 (0.514) | -0.304 (0.516)

7. Secondary Outcome: Change From Baseline in the Mean Plasma D-serine to Total Serine Ratio at Day 8
Description: Blood samples were collected at pre-specified timepoints and plasma concentrations of D-serine and total serine were measured. Plasma D-serine to total serine ratios were then calculated. Results are reported as LS mean change from baseline at Day 8, determined using a MMRM.
Time Frame: Baseline and Day 8 of each treatment period
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Luvadaxistat 50 mg | Placebo (Reference for Luvadaxistat 50 mg) | Luvadaxistat 500 mg | Placebo (Reference for Luvadaxistat 500 mg)
Number analyzed (Participants) | 12 | 12 | 15 | 15
ratio | 0.00293 (0.000855) | 0.000590 (0.000863) | 0.00561 (0.000994) | 0.000620 (0.000997)

8. Secondary Outcome: Mean Plasma Concentration of Luvadaxistat
Description: Blood samples were collected at pre-specified timepoints and plasma concentrations of luvadaxistat were measured.
Time Frame: Day 1 0.25 to 2 hours and 3 to 6 hours post-dose, Day 7 pre-dose, 0.25 to 2 hours and 3 to 6 hours post-dose, and Day 8 pre-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanograms / milliliter
Arm/Group | Luvadaxistat 50 mg | Luvadaxistat 500 mg
Number analyzed (Participants) | 14 | 15
nanograms / milliliter
  Day 1 - Post-dose (0.25 to 2 hours) | 253.4 (199.3) | 700.4 (783.0)
  Day 1 - Post-dose (3 to 6 hours) | 47.66 (35.64) | 671.1 (473.1)
  Day 7 - Pre-dose | 8.749 (19.212) | 78.92 (229.90)
  Day 7 - Post-dose (0.25 to 2 hours): number analyzed (Participants) | 13 | 15
  Day 7 - Post-dose (0.25 to 2 hours) | 203.5 (199.6) | 1184 (482)
  Day 7 - Post-dose (3 to 6 hours): number analyzed (Participants) | 13 | 15
  Day 7 - Post-dose (3 to 6 hours) | 38.94 (26.23) | 301.5 (177.2)
  Day 8 - Pre-dose: number analyzed (Participants) | 12 | 15
  Day 8 - Pre-dose | 3.366 (2.726) | 21.61 (14.65)

ADVERSE EVENTS:
Time Frame: 8-day treatment period for each of treatment periods 1 and 2 (separated by washout of up to 21 days) and up to 30 days follow-up after last dose of study treatment. Up to a maximum of 67 days for overall timeframe.
Description: Treatment-emergent adverse events were defined as adverse events that occurred after the first dose of study treatment and up to 30 days after the last dose or early termination. The safety analysis set included all randomized participants who received at least 1 dose of study treatment.
Groups:
- Placebo: Participants who received matching placebo orally QD for 8 days during either treatment periods 1 or 2 of the study. Placebo treatment was pooled for participants receiving 50 mg and 500 mg luvadaxistat.
Arm/Group | Placebo | Luvadaxistat 500 mg | Luvadaxistat 50 mg
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/29 | 0/15 | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=29) | Luvadaxistat 500 mg (N=15) | Luvadaxistat 50 mg (N=14)
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-01-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT03359785/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/85/NCT03359785/SAP_001.pdf